CLINICAL TRIAL: NCT03998865
Title: Bacterial Microbiota and Its Relation to Antimicrobial Resistance Genes in Implant-supported PEEK and Titanium Provisional Abutments
Brief Title: Bacterial Microbiota Characterization on Implant-supported PEEK and Titanium Provisional Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Wendler Ernst (Other)
Responsible Party: Sponsor-Investigator, Michael Wendler Ernst, Assistant Professor at the Department of Restorative Dentistry, Faculty of Dentistry, University of Concepcion, Chile
Organization: University of Concepcion, Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 218.102.032-1.0IN
Record Dates: First submitted 2019-06-12; First posted 2019-06-26 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Peri-implant Mucositis; Oral Bacterial Infection; Bacterial Resistance
Keywords: Implant-supported Provisional Abutment; Poly-ether-ether-ketone; Titanium; Bacterial Microbiota; Antimicrobial Resistance Genes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: PEEK or Titanium provisional-abutments. A sample of the niche microbiota will be retrieved prior to implant placement (t0) and two months after provisional abutment (crown) connection (t1).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be not aware of the type of provisional abutment used in their treatment. Retrieved samples will be codified in order to mask them for the metagenomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK Provisional Abutment (Experimental): The provisional crown will be fixed onto a PEEK abutment and then connected to the implant. The bis-acrylic resin used for the provisional crown will not invade the emergence profile of the abutment.
  Interventions: Device: Provisional abutment material
- Titanium Provisional Abutment (Active Comparator): The provisional crown will be fixed onto a titanium abutment and then connected to the implant. The bis-acrylic resin used for the provisional crown will not invade the emergence profile of the abutment.
  Interventions: Device: Provisional abutment material

INTERVENTIONS:
Device: Provisional abutment material — The effect of the provisional abutment material on the characteristics of the bacterial microbiota will be assessed by using PEEK (experimental) or Titanium (active comparator) provisional abutments.

SUMMARY:
The aim of this study is to determine the relative abundances of the different bacterial phyla and families in the microbiota present on the surface of PEEK implant-supported provisional abutments compared to titanium implant-supported provisional abutments, as well as the effect of both materials on the presence of antibiotics resistance genes.

DETAILED DESCRIPTION:
The use of provisional abutments is mandatory during the restorative phase of any implant based oral rehabilitation. The introduction of poly-ether-ether-ketone (PEEK) for the manufacturing of provisional abutments as an alternative to conventional titanium abutments has opened the restorative spectra, offering the clinician and the patient better aesthetics and adhesive outcomes than its predecessor. However, there is to date no clarity on the impact of PEEK on the bacterial growth and the specificity of the microbiota on the abutment surface. Therefore, the present study aims to determine the relative abundances of the different bacterial phyla and families in the microbiota present on the surface of PEEK and titanium implant-supported provisional abutments, as well as the effect of both materials on the presence of antibiotics resistance genes.

Study Hypotheses:

* H1: The characteristics of the bacterial microbiota present at the connection area of implant-supported provisional abutments are dependent upon the abutment material.
* H2: An increased presence of antibiotic resistance genes is found in the bacterial microbiota on titanium provisional abutments when compared to that found on PEEK abutments.

The study uses a metagenomic approach based on the characterization of the bacterial communities, as well as on the sequencing of the 16S gene, and on the other hand, on the sequencing of the high-throughput (HTS) of the whole genome, for variations of the antibiotic resistance genes.

Sample retrieval will be conducted prior to implant placement, at the adjacent teeth gingival sulcus (t0), and two months after provisional abutment (and crown) connection (t1), from the retrieved abutments. Patient allocation in the "PEEK" or "Titanium" groups will be randomized. Intra- and interpatient comparisons will be conducted. Statistical analyses include two-way ANOVA and Tukey's post-hoc test, at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* ASA I patients
* Indication of implant treatment to replace an upper or lower premolar
* Presence of natural teeth adjacent to the implant region
* Gingival biotype in the posterior region of 3 to 4 mm

Exclusion Criteria:

* Immunosuppressed patients
* Tabacco, alcohol or drug addictions
* History of periodontal disease
* Need of bone grafting in the implant region

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in the Number of Operational Taxonomic Units (OTUS) | Baseline (prior to abutment insertion) and two months after abutment insertion.
  Changes in the Number of Operational Taxonomic Units (OTUS) observed after the two months evaluation period will be assessed using UniFrac metrics. The weighted UniFrac distances will be used to perform a principal coordinate analysis (PCO).
Changes in Antibacterial Resistance Genes (ARG) | Baseline (prior to abutment insertion) and two months after abutment insertion.
  Changes in the ARG of the microbiota will be determined using the whole genome sequencing using the MiSeq Illumina method.

SECONDARY OUTCOMES:
Changes in the number of bacterial species | Baseline (prior to abutment insertion) and two months after abutment insertion.
  Changes in the bacterial microbiota richness will be evaluated using a bias corrected Chao 1 richness estimator and the Shannon diversity index.

CONTACTS AND LOCATIONS:
Overall Officials: Michael U Wendler, DDS, PhD, Principal Investigator — Department of Restorative Dentistry, University of Concepcion
Locations (1):
- Department of Restorative Dentistry, Faculty of Dentistry, University of Concepcion, Concepción, Bio Bio, Chile

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be communicated, in accordance with the ethical approval of the study. Data will be communicated grouped with the individual effects on the results assessed with the respective statistical tools.

REFERENCES:
- [Background] Schwitalla AD, Abou-Emara M, Zimmermann T, Spintig T, Beuer F, Lackmann J, Muller WD. The applicability of PEEK-based abutment screws. J Mech Behav Biomed Mater. 2016 Oct;63:244-251. doi: 10.1016/j.jmbbm.2016.06.024. Epub 2016 Jul 1. PMID 27434650
- [Background] Mawhinney J, Connolly E, Claffey N, Moran G, Polyzois I. An in vivo comparison of internal bacterial colonization in two dental implant systems: identification of a pathogenic reservoir. Acta Odontol Scand. 2015 Apr;73(3):188-94. doi: 10.3109/00016357.2014.978365. Epub 2014 Nov 11. PMID 25385682
- [Background] Barbosa RE, do Nascimento C, Issa JP, Watanabe E, Ito IY, de Albuquerque RF Jr. Bacterial culture and DNA Checkerboard for the detection of internal contamination in dental implants. J Prosthodont. 2009 Jul;18(5):376-81. doi: 10.1111/j.1532-849X.2009.00454.x. Epub 2009 Apr 3. PMID 19374709
- [Background] Broggini N, McManus LM, Hermann JS, Medina RU, Oates TW, Schenk RK, Buser D, Mellonig JT, Cochran DL. Persistent acute inflammation at the implant-abutment interface. J Dent Res. 2003 Mar;82(3):232-7. doi: 10.1177/154405910308200316. PMID 12598555
- [Background] Subramani K, Jung RE, Molenberg A, Hammerle CH. Biofilm on dental implants: a review of the literature. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):616-26. PMID 19885401
- [Background] Campoccia D, Montanaro L, Arciola CR. The significance of infection related to orthopedic devices and issues of antibiotic resistance. Biomaterials. 2006 Apr;27(11):2331-9. doi: 10.1016/j.biomaterials.2005.11.044. Epub 2005 Dec 20. PMID 16364434
- [Background] Romanos GE, Biltucci MT, Kokaras A, Paster BJ. Bacterial Composition at the Implant-Abutment Connection under Loading in vivo. Clin Implant Dent Relat Res. 2016 Feb;18(1):138-45. doi: 10.1111/cid.12270. Epub 2014 Sep 5. PMID 25195711
- [Background] Weber DJ, Rutala WA. Self-disinfecting surfaces: review of current methodologies and future prospects. Am J Infect Control. 2013 May;41(5 Suppl):S31-5. doi: 10.1016/j.ajic.2012.12.005. PMID 23622745
- [Background] Baker-Austin C, Wright MS, Stepanauskas R, McArthur JV. Co-selection of antibiotic and metal resistance. Trends Microbiol. 2006 Apr;14(4):176-82. doi: 10.1016/j.tim.2006.02.006. Epub 2006 Mar 14. PMID 16537105
- [Background] Di Cello F, Pepi M, Baldi F, Fani R. Molecular characterization of an n-alkane-degrading bacterial community and identification of a new species, Acinetobacter venetianus. Res Microbiol. 1997 Mar-Apr;148(3):237-49. doi: 10.1016/S0923-2508(97)85244-8. PMID 9765804
- [Background] Diaz PI, Dupuy AK, Abusleme L, Reese B, Obergfell C, Choquette L, Dongari-Bagtzoglou A, Peterson DE, Terzi E, Strausbaugh LD. Using high throughput sequencing to explore the biodiversity in oral bacterial communities. Mol Oral Microbiol. 2012 Jun;27(3):182-201. doi: 10.1111/j.2041-1014.2012.00642.x. Epub 2012 Mar 3. PMID 22520388
- [Background] Sanchez-Sanhueza G, Bello-Toledo H, Gonzalez-Rocha G, Goncalves AT, Valenzuela V, Gallardo-Escarate C. Metagenomic study of bacterial microbiota in persistent endodontic infections using Next-generation sequencing. Int Endod J. 2018 Dec;51(12):1336-1348. doi: 10.1111/iej.12953. Epub 2018 Jun 9. PMID 29786880